CLINICAL TRIAL: NCT00860847
Title: Firefighter Aged Garlic Extract Investigation With CoQ10 as a Treatment for Heart Disease (FAITH)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Responsible Party: Principal Investigator, Matthew J. Budoff, Professor of Medicine, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Wakunaga of America Co., Ltd.
Record Dates: First submitted 2009-03-11; First posted 2009-03-12 (Estimated); Results first posted 2015-03-12 (Estimated); Last update posted 2015-03-12 (Estimated); Status verified 2015-02

CONDITIONS: Coronary Atherosclerosis; Coronary Artery Calcification; Coronary Stenosis
Keywords: Progression of Atherosclerosis; Aged garlic extract; Biomarkers of inflammation; Coronary Plaque Volume and coronary Stenosis; Vascular function
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis | interventions — coenzyme Q10

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aged Garlic Extract and Coenzyme Q10 (Active Comparator): AGE (1200 mg) and CoQ10 (120 mg)
  This is a combination of aged garlic extract and co-enzyme Q10
  Interventions: Dietary Supplement: Aged garlic extract and Coenzyme Q10
- Placebo (No Intervention): placebo pills will be given

INTERVENTIONS:
Dietary Supplement: Aged garlic extract and Coenzyme Q10 — AGE (1200 mg) and CoQ10 (120 mg)
  Other Names: Kyolic formula 110
  Arms: Aged Garlic Extract and Coenzyme Q10

SUMMARY:
1. Statement of Problem

   According to the National Fire Protection Association (NFPA), 43.7% of all firefighters that died on the job experienced sudden cardiac death. The job also affords an incredible amount of stress. Cholesterol therapy has been well demonstrated to reduce coronary plaque progression. However is certainly not the only factor in evaluating for progression of coronary artery disease (CAD), and other factors must play a role. Garlic therapy has been shown to retard atherosclerosis independently.
2. Hypothesis and Specific Aims The hypothesis of this proposal is: In comparison to the placebo group, Aged Garlic Extract (AGE) therapy + Coenzyme Q10 (CoQ10) will be effective in slowing progression of coronary artery calcification (CAC) in firefighters with established atherosclerosis, independent of baseline blood pressure, statin use or other cardiovascular risk factors.

Specific Aims:

1. Compare the effects of cholesterol lowering effects in a firefighter population of patients under the influence of Aged Garlic Extract + CoQ10 or placebo.
2. Compare whether degree of change in atherosclerotic coronary artery plaque burden will change at a different rate under the influence of Aged Garlic Extract + CoQ10 compared to placebo treatment.
3. Compare whether Aged Garlic Extract + CoQ10 therapy induces changes in baseline values including biological and biochemical parameters, such as LDL cholesterol, homocysteine, C-reactive protein (CRP), and endothelial function.

DETAILED DESCRIPTION:
Inclusion Criteria

* Calcium scan with Agatston score >20
* Age 35-84 years
* Subjects must provide written informed consent after the scope and nature of the investigation has been explained to them
* Subjects should be stable on their concomitant medications for at least 12 weeks prior to randomization
* Subjects who agree to refrain from supplemental garlic or significant dietary garlic

Exclusion Criteria

* A contraindication to Aged Garlic Extract therapy including: known hypersensitivity to drug.
* Any unstable medical, psychiatric or substance abuse disorder that in the opinion of the investigator or principal investigator is likely to affect the subject's ability to complete the study or precludes the subject's participation in the study
* Weight in excess of 325 pounds
* Bleeding disorder
* History of myocardial infarction, stroke or life-threatening arrhythmia within the prior six months
* Resting hypotension (a resting systolic blood pressure of <90 mm Hg) or hypertension (a resting blood pressure > 170 mm Hg or a resting diastolic blood pressure of >110 mm Hg)
* NYHA Class III or IV heart failure
* History of malignancy within the last 5 years (other than skin cancer) or evidence of active cancer which would require concomitant cancer chemotherapy
* Serum creatinine > 1.4 mg/dl
* Triglycerides > 400 at visit 1
* Diabetic subjects with HbA1c > 12%
* Drug or alcohol abuse, or current intake of more than 14 standard drinks per week
* Concurrent enrollment in another placebo-controlled trial
* Presence of metal clips (i.e. bypass patients) or intracoronary stenting that preclude accurate measure of coronary calcification
* Partial ileal bypass or known gastrointestinal disease limiting drug absorption
* Current intake of garlic supplement or other prohibited drug (Appendix B)
* Current tobacco use
* Current use of anticoagulants (except for antiplatelet agents)
* Chronic renal failure
* Hematological or biochemical values at screening outside the reference ranges considered as clinically significant in the opinion of the investigator or PI

Outcome Measures Primary - Rate of change in total coronary calcium scores by CT The Agatston score was calculated by multiplying the lesion area (mm^2) by a density factor. The density was measured in Hounsfield units, and score of 1 for 130-199 HU, 2 for 200-299 HU, 3 for 300-399 HU, and 4 for 400 HU and greater.

Secondary Change in blood values and endothelial function over 6 and 12 months:

1. Plasma lipids: total plasma cholesterol and triglycerides, LDL-Cholesterol, HDL-Cholesterol, and VLDL-Cholesterol determined by the precipitation method;
2. Endothelial markers and inflammation: C-reactive protein and Homocysteine, as well as GSH

ELIGIBILITY:
Inclusion Criteria:

* Calcium scan with Agatston score >20
* Age 35-84 years
* Subjects must provide written informed consent after the scope and nature of the investigation has been explained to them
* Subjects should be stable on their concomitant medications for at least 12 weeks prior to randomization
* Subjects who agree to refrain from supplemental garlic or significant dietary garlic

Exclusion Criteria:

* A contraindication to Aged Garlic Extract therapy including: known hypersensitivity to drug.
* Any unstable medical, psychiatric or substance abuse disorder that in the opinion of the investigator or principal investigator is likely to affect the subject's ability to complete the study or precludes the subject's participation in the study
* Weight in excess of 325 pounds
* Bleeding disorder
* History of myocardial infarction, stroke or life-threatening arrhythmia within the prior six months
* Resting hypotension (a resting systolic blood pressure of <90 mm Hg) or hypertension (a resting blood pressure > 170 mm Hg or a resting diastolic blood pressure of >110 mm Hg)
* NYHA Class III or IV heart failure
* History of malignancy within the last 5 years (other than skin cancer) or evidence of active cancer which would require concomitant cancer chemotherapy
* Serum creatinine > 1.4 mg/dl
* Triglycerides > 400 at visit 1
* Diabetic subjects with HbA1c > 12%
* Drug or alcohol abuse, or current intake of more than 14 standard drinks per week
* Concurrent enrollment in another placebo-controlled trial
* Presence of metal clips (i.e. bypass patients) or intracoronary stenting that preclude accurate measure of coronary calcification
* Partial ileal bypass or known gastrointestinal disease limiting drug absorption
* Current intake of garlic supplement or other prohibited drug (Appendix B)
* Current tobacco use
* Current use of anticoagulants (except for antiplatelet agents)
* Chronic renal failure
* Hematological or biochemical values at screening outside the reference ranges considered as clinically significant in the opinion of the investigator or PI

Ages: 35 Years to 84 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2009-05; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Budoff, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Los Angeles Biomedical Research Institute, Torrance, California, United States

REFERENCES:
- [Background] Libby P, Schoenbeck U, Mach F, Selwyn AP, Ganz P. Current concepts in cardiovascular pathology: the role of LDL cholesterol in plaque rupture and stabilization. Am J Med. 1998 Feb 23;104(2A):14S-18S. doi: 10.1016/s0002-9343(98)00041-2. PMID 9550502
- [Background] Lau BH, Li L, Yoon P. Thymic peptide protects vascular endothelial cells from hydrogen peroxide-induced oxidant injury. Life Sci. 1993;52(22):1787-96. doi: 10.1016/0024-3205(93)90468-i. PMID 8492641
- [Background] Weissberg PL, Bennett MR. Atherosclerosis--an inflammatory disease. N Engl J Med. 1999 Jun 17;340(24):1928-9. No abstract available. PMID 10375320
- [Background] Raggi P, Callister TQ, Shaw LJ. Progression of coronary artery calcium and risk of first myocardial infarction in patients receiving cholesterol-lowering therapy. Arterioscler Thromb Vasc Biol. 2004 Jul;24(7):1272-7. doi: 10.1161/01.ATV.0000127024.40516.ef. Epub 2004 Apr 1. PMID 15059806
- [Background] Budoff MJ, Takasu J, Flores FR, Niihara Y, Lu B, Lau BH, Rosen RT, Amagase H. Inhibiting progression of coronary calcification using Aged Garlic Extract in patients receiving statin therapy: a preliminary study. Prev Med. 2004 Nov;39(5):985-91. doi: 10.1016/j.ypmed.2004.04.012. PMID 15475033
- [Background] Steiner M, Lin RS. Changes in platelet function and susceptibility of lipoproteins to oxidation associated with administration of aged garlic extract. J Cardiovasc Pharmacol. 1998 Jun;31(6):904-8. doi: 10.1097/00005344-199806000-00014. PMID 9641475
- [Background] BEUTLER E, DURON O, KELLY BM. Improved method for the determination of blood glutathione. J Lab Clin Med. 1963 May;61:882-8. No abstract available. PMID 13967893
- [Background] Mao S, Bakhsheshi H, Lu B, Liu SC, Oudiz RJ, Budoff MJ. Effect of electrocardiogram triggering on reproducibility of coronary artery calcium scoring. Radiology. 2001 Sep;220(3):707-11. doi: 10.1148/radiol.2203001129. PMID 11526270
- [Background] Ahmadi N, Hajsadeghi F, Gul K, Vane J, Usman N, Flores F, Nasir K, Hecht H, Naghavi M, Budoff M. Relations between digital thermal monitoring of vascular function, the Framingham risk score, and coronary artery calcium score. J Cardiovasc Comput Tomogr. 2008 Nov;2(6):382-8. doi: 10.1016/j.jcct.2008.09.001. Epub 2008 Sep 26. PMID 19083982

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 65 patients were recruited
Pre-assignment Details: completed
Groups:
- Aged Garlic Extract and Coenzyme Q10: Patients randomized to oral AGE (1200 mg) and CoQ10 (120 mg)
- Placebo: Patients randomized to placebo
Period: Overall Study
Arm/Group | Aged Garlic Extract and Coenzyme Q10 | Placebo
Started | 32 | 33
Completed | 28 | 28
Not Completed | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aged Garlic Extract and Coenzyme Q10 | Placebo | Total
Number analyzed (Participants) | 32 | 33 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 33 | 65
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (6) | 55 (6) | 55 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 17 | 17 | 34
Region of Enrollment [Number; unit: participants]
  United States | 32 | 33 | 65

OUTCOME MEASURES:

1. Primary Outcome: Rate of Change in Total Coronary Calcium Scores by Computed Tomography
Description: progression of coronary artery calcium deposits as determined by computed tomography as measured by the Agatston score: The Agatston score was calculated by multiplying the lesion area (mm^2) by a density factor. The density was measured in Hounsfield units, and score of 1 for 130-199 HU, 2 for 200-299 HU, 3 for 300-399 HU, and 4 for 400 HU and greater The endpoint is the mean change (end of study value - baseline value) in each group.
Time Frame: 1 year
Population: all participants were analyzed
Measure: Mean (Standard Deviation); unit: Agatston score change
Arm/Group | Aged Garlic Extract and Coenzyme Q10 | Placebo
Number analyzed (Participants) | 32 | 33
Agatston score change | 32 (6) | 58 (8)

2. Secondary Outcome: 1.Plasma Lipids: Total Plasma Cholesterol and Triglycerides, LDL-Cholesterol, HDL-Cholesterol, and VLDL-Cholesterol Determined by the Precipitation Method; 2. Endothelial Markers and Inflammation: C-reactive Protein and Homocysteine, as Well as GSH
Time Frame: 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Aged Garlic Extract and Coenzyme Q10 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/33
Other Adverse Events (participants affected / at risk) | 0/32 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No